CLINICAL TRIAL: NCT04679285
Title: Pilot Study to Assess Minimal Residual Disease on Cryopreserved Ovarian Fragments in Younger Patients Treated for Acute Myeloid Leukemia
Brief Title: Minimal Residual Disease Evaluation on Cryopreserved Ovarian Fragments in Younger Patients Treated for Acute Myeloid Leukemia
Acronym: FERTILAM
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Canceropôle Nord Ouest (Other); Saint-Louis Hospital, Paris, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_12; 2020-A01513-36 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-12-16; First posted 2020-12-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; Fertility preservation; Ovarian cryopreservation; Minimal residual disease
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Bone marrow, blood, ovarian fragments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cryopreservation of ovarian cortex represents an option for fertility preservation in patients diagnosed with acute myeloid leukemia and requiring allogeneic stem cell transplantation.

This pilot study aims to evaluate the minimal residual disease on ovarian fragments harvested before allogeneic stem cell transplantation at the time of complete remission.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with AML
* At least one molecular marker identified at AML diagnosis
* Patients who undergo ovarian tissue cryopreservation for fertility preservation in complete remission, before hematopoietic stem cell transplantation.

Exclusion Criteria:

* Other diagnostic
* No marker available at AML diagnosis
* No bone marrow/ovarian fragment available at the time of complete remission

Ages: 2 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Patients aged 2 to 40 year-old, who present at least one molecular marker at acute myeloid leukemia diagnosis and who undergo ovarian cryopreservation for fertility preservation at the time of complete remission, before hematopoietic stem cell transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-09-04 (Actual); Study Completion 2022-09-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patients without detectable MRD in ovarian tissue | Up to 6 months

SECONDARY OUTCOMES:
Percentage of patients with MRD detected in ovarian tissue and bone marrow. | Up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Laurène Fenwarth, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU lille, Lille, France